CLINICAL TRIAL: NCT04053452
Title: Peripheral Nerve Ultrasound for Diagnosis and Prognosis of Guillain-Barre Syndrome: A Pilot Study
Brief Title: Peripheral Nerve Ultrasound for Diagnosis and Prognosis of Guillain-Barre Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Duke University (Other)
Collaborators: GBS-CIDP foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00102385
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-03

CONDITIONS: Guillain-Barre Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The EMG lab physician or technician performing the ultrasound will be blinded to the EMG/NCS results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- GBS Patients (Experimental)
  Interventions: Diagnostic Test: Peripheral nerve ultrasound; Diagnostic Test: Measurement of strength
- Controls (Active Comparator)
  Interventions: Diagnostic Test: Peripheral nerve ultrasound

INTERVENTIONS:
Diagnostic Test: Peripheral nerve ultrasound — Ultrasound of the bilateral ulnar nerves, median nerves, vagus nerves, and C6 and C7 nerve roots will be performed.
Diagnostic Test: Measurement of strength — Strength will be assessed by physical examination and recorded using Medical Research Council (MRC) scale, and a hand dynamometer will be used to measure grip strength.
  Arms: GBS Patients

SUMMARY:
The purpose of this study is to determine if peripheral nerve ultrasound can be used as a supplemental tool to diagnose Guillain-Barre syndrome (GBS) in the acute setting and aid in prognostication.

ELIGIBILITY:
Inclusion Criteria:

* For GBS group: Inpatients with acute, progressive weakness and no alternative diagnosis, with onset less than 30 days prior to examination.
* For control group: Hospitalized patients on the inpatient neurology service who are being treated for non-peripheral nerve disorders (e.g. epilepsy, multiple sclerosis, or stroke).
* For all subjects: 18+ years of age

Exclusion Criteria:

- Patients with any history of multifocal motor neuropathy (MMN), prior Guillain-Barre syndrome (GBS), chronic inflammatory demyelinating polyneuropathy (CIDP), or hereditary neuropathy (e.g. Charcot-Marie-Tooth)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2024-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hobson-Webb, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GBS Patients | Controls
Started | 14 | 6
Completed | 12 | 4
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Time restraint due to inpatient needs | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GBS Patients | Controls | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.71 (13.93) | 59.30 (15.19) | 58.23 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 8 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 13 | 5 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Internerve Variability of Cross-sectional Area (CSA) in Patients With GBS vs Controls
Description: Internerve CSA variability for each patient will be calculated as: maximal intranerve CSA variability/minimal intranerve CSA variability. Intranerve CSA variability for each nerve will be calculated as: maximal CSA/minimal CSA for median and ulnar nerves.
Time Frame: Day 0 and approximately 7 days after admission
Population: Participants with data collected at each time point.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | GBS Patients | Controls
Number analyzed (Participants) | 14 | 6
mm^2
  Day 0 | 1.82 (0.43) | 1.49 (0.31)
  Day 7: number analyzed (Participants) | 1 | 0
  Day 7 | 1.38 (0) |
Statistical Analysis 1: Comparison: GBS Patients vs Controls; Test type: Other; Area under the curve = 0.7262 — Area under the receiver operating characteristic (ROC) curve

2. Primary Outcome: Median Nerve Intranerve Cross-sectional Area (CSA) Variability in Patients With GBS vs Controls
Description: Intranerve CSA variability for each nerve is calculated as: maximal intranerve CSA/minimal intranerve CSA . When both left and right ulnar nerves were scanned, the side with the largest intranerve CSA variability was used for analysis.
Time Frame: Day 0 and approximately 7 days after admission
Population: Participants with data collected at each time point.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | GBS Patients | Controls
Number analyzed (Participants) | 14 | 6
mm^2
  Day 0 | 1.96 (0.51) | 1.73 (0.56)
  Day 7: number analyzed (Participants) | 1 | 0
  Day 7 | 1.63 (0) |
Statistical Analysis 1: Comparison: GBS Patients vs Controls; Test type: Other; Area under the curve = 0.6667 — Area under the receiver operating characteristic (ROC) curve

3. Primary Outcome: Ulnar Nerve Intranerve Cross-sectional Area (CSA) Variability in Patients With GBS vs Controls
Description: as for outcome 2
Time Frame: Day 0 and approximately 7 days after admission
Population: Participants with data collected at each time point.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | GBS Patients | Controls
Number analyzed (Participants) | 14 | 6
mm^2
  Day 0 | 2.36 (0.71) | 1.88 (0.65)
  Day 7: number analyzed (Participants) | 1 | 0
  Day 7 | 2.25 (0) |
Statistical Analysis 1: Comparison: GBS Patients vs Controls; Test type: Other; Area under the curve = 0.7083 — Area under the receiver operating characteristic (ROC) curve

4. Secondary Outcome: Length of Hospital Stay in Days
Description: Length of hospital stay is measured to the nearest day (by chart review).
Time Frame: Up to approximately 20 days
Population: Not applicable to the Control group.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GBS Patients | Controls
Number analyzed (Participants) | 14 | 0
days | 12.93 (6.21) |
Statistical Analysis 1: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Median at wrist; Kendall's tau correlation coefficient = -0.0623, 95% CI 2-sided [-0.5005 to 0.4791]
Statistical Analysis 2: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Median at forearm; Kendall's tau correlation coefficient = -0.1628, 95% CI 2-sided [-0.6503 to 0.4222]
Statistical Analysis 3: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Median at cubital fossa; Kendall's tau correlation coefficient = -0.1850, 95% CI 2-sided [-0.5490 to 0.1829]
Statistical Analysis 4: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Median at humerus; Kendall's tau correlation coefficient = 0.0512, 95% CI 2-sided [-0.3411 to 0.5017]
Statistical Analysis 5: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Median at axilla; Kendall's tau correlation coefficient = 0.0476, 95% CI 2-sided [-0.4335 to 0.5592]
Statistical Analysis 6: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Ulnar at wrist; Kendall's tau correlation coefficient = -0.1229, 95% CI 2-sided [-0.5092 to 0.3040]
Statistical Analysis 7: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Ulnar at forearm; Kendall's tau correlation coefficient = 0.0603, 95% CI 2-sided [-0.3057 to 0.4137]
Statistical Analysis 8: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Ulnar at cubital fossa; Kendall's tau correlation coefficient = 0.1059, 95% CI 2-sided [-0.4028 to 0.5700]
Statistical Analysis 9: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Ulnar at humerus; Kendall's tau correlation coefficient = -0.1786, 95% CI 2-sided [-0.6503 to 0.2838]
Statistical Analysis 10: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Ulnar at axilla; Kendall's tau correlation coefficient = -0.2396, 95% CI 2-sided [-0.5714 to 0.1950]
Statistical Analysis 11: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — C6; Kendall's tau correlation coefficient = -0.0671, 95% CI 2-sided [-0.4667 to 0.3336]
Statistical Analysis 12: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — C7; Kendall's tau correlation coefficient = -0.2134, 95% CI 2-sided [-0.7018 to 0.3193]
Statistical Analysis 13: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and length of hospital stay; Test type: Other — Vagus; Kendall's tau correlation coefficient = 0.0246, 95% CI 2-sided [-0.3506 to 0.4596]

5. Secondary Outcome: Ambulatory Status on Discharge
Description: Number of participants with ambulatory status as "ambulatory with or without assistance".
Time Frame: At discharge, up to approximately 20 days
Population: Not applicable to the Control group.
Measure: Count of Participants; unit: Participants
Arm/Group | GBS Patients | Controls
Number analyzed (Participants) | 14 | 0
Participants | 6 |
Statistical Analysis 1: Comparison: GBS Patients; Null hypothesis: Nerve ultrasound measurement has no effect on the log-odds of walking (i.e., nerve ultrasound measurements do not predict whether a subject is ambulatory at discharge); Test type: Other — Median at wrist; p = 0.360, Regression, Logistic; Odds Ratio (OR) = 0.7686494
Statistical Analysis 2: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — Median at forearm; p = 0.521, Regression, Logistic; Odds Ratio (OR) = 0.9315228
Statistical Analysis 3: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — Median at cubital fossa; p = 0.245, Regression, Logistic; Odds Ratio (OR) = 0.7949528
Statistical Analysis 4: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — Median at humerus; p = 0.541, Regression, Logistic; Odds Ratio (OR) = 0.8603349
Statistical Analysis 5: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — Median at axilla; p = 0.415, Regression, Logistic; Odds Ratio (OR) = 0.8767973
Statistical Analysis 6: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — Ulnar at wrist; p = 0.504, Regression, Logistic; Odds Ratio, log = 0.7613965
Statistical Analysis 7: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — Ulnar at forearm; p = 0.393, Regression, Logistic; Odds Ratio (OR) = 0.8061505
Statistical Analysis 8: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — Ulnar at cubital fossa; p = 0.222, Regression, Logistic; Odds Ratio (OR) = 0.8336885
Statistical Analysis 9: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — Ulnar at humerus; p = 0.615, Regression, Logistic; Odds Ratio (OR) = 1.1214848
Statistical Analysis 10: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — Ulnar at axilla; p = 0.926, Regression, Logistic; Odds Ratio (OR) = 0.9898411
Statistical Analysis 11: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — C6; p = 0.519, Regression, Logistic; Odds Ratio (OR) = 0.9402829
Statistical Analysis 12: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — C7; p = 0.379, Regression, Logistic; Odds Ratio (OR) = 0.9347906
Statistical Analysis 13: Comparison: GBS Patients; [analysis description as in outcome 5, analysis 1]; Test type: Other — Vagus; p = 0.511, Regression, Logistic; Odds Ratio (OR) = 0.8968658

6. Secondary Outcome: Respiratory Dysfunction, as Measured by Number of Days Intubated
Description: Respiratory dysfunction will be measured by number of days intubated (to the nearest day) by chart review.
Time Frame: During admission, up to approximately 20 days
Population: Not applicable to the Control group.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GBS Patients | Controls
Number analyzed (Participants) | 14 | 0
days | 1.29 (3.00) |
Statistical Analysis 1: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Median at wrist; Kendall's tau correlation coefficient = -0.0577350, 95% CI 2-sided [-0.4273 to 0.3293]
Statistical Analysis 2: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Median at forearm; Kendall's tau correlation coefficient = -0.0359442, 95% CI 2-sided [-0.5480 to 0.5248]
Statistical Analysis 3: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Median at cubital fossa; Kendall's tau correlation coefficient = 0.1429483, 95% CI 2-sided [-0.1938 to 0.4763]
Statistical Analysis 4: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Median at humerus; Kendall's tau correlation coefficient = -0.3955939, 95% CI 2-sided [-0.6811 to -0.0874]
Statistical Analysis 5: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Median at axilla; Kendall's tau correlation coefficient = -0.3681051, 95% CI 2-sided [-0.7032 to 0.1185]
Statistical Analysis 6: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Ulnar at wrist; Kendall's tau correlation coefficient = -0.4938292, 95% CI 2-sided [-0.7112 to -0.1978]
Statistical Analysis 7: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Ulnar at forearm; Kendall's tau correlation coefficient = 0.1304373, 95% CI 2-sided [-0.2201 to 0.5014]
Statistical Analysis 8: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Ulnar at cubital fossa; Kendall's tau correlation coefficient = 0.3273268, 95% CI 2-sided [-0.0679 to 0.6612]
Statistical Analysis 9: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Ulnar at humerus; Kendall's tau correlation coefficient = -0.0552157, 95% CI 2-sided [-0.4213 to 0.3610]
Statistical Analysis 10: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Ulnar at axilla; Kendall's tau correlation coefficient = -0.1666667, 95% CI 2-sided [-0.5389 to 0.2057]
Statistical Analysis 11: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — C6; Kendall's tau correlation coefficient = -0.3194892, 95% CI 2-sided [-0.6539 to 0.2288]
Statistical Analysis 12: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — C7; Kendall's tau correlation coefficient = -0.4959498, 95% CI 2-sided [-0.6860 to -0.2065]
Statistical Analysis 13: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and respiratory dysfunction; Test type: Other — Vagus; Kendall's tau correlation coefficient = -0.3228883, 95% CI 2-sided [-0.6487 to 0.0000]

7. Secondary Outcome: Strength, as Measured by Hand Dynamometer
Description: Average of left and right hand grip strength (in pounds).
Time Frame: Day 0, Day 7
Population: Participants with data collected at each time point. Not applicable to the Control group.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | GBS Patients | Controls
Number analyzed (Participants) | 13 | 0
lbs
  Day 0 | 37.17 (25.37) |
  Day 7: number analyzed (Participants) | 1 | 0
  Day 7 | 80.00 (0) |
Statistical Analysis 1: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Median at wrist; Kendall's tau correlation coefficient = -0.1415346, 95% CI 2-sided [-0.7350 to 0.4247]
Statistical Analysis 2: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Median at forearm; Kendall's tau correlation coefficient = 0.1987845, 95% CI 2-sided [-0.4377 to 0.8004]
Statistical Analysis 3: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Median at cubital fossa; Kendall's tau correlation coefficient = -0.0789747, 95% CI 2-sided [-0.5256 to 0.3778]
Statistical Analysis 4: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Median at humerus; Kendall's tau correlation coefficient = 0.1621509, 95% CI 2-sided [-0.3591 to 0.5606]
Statistical Analysis 5: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Median at axilla; Kendall's tau correlation coefficient = 0.1499412, 95% CI 2-sided [-0.3901 to 0.6374]
Statistical Analysis 6: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Ulnar at wrist; Kendall's tau correlation coefficient = -0.0140441, 95% CI 2-sided [-0.5773 to 0.5407]
Statistical Analysis 7: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Ulnar at forearm; Kendall's tau correlation coefficient = 0.01383297, 95% CI 2-sided [-0.5288 to 0.5485]
Statistical Analysis 8: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Ulnar at cubital fossa; Kendall's tau correlation coefficient = -0.2935683, 95% CI 2-sided [-0.6968 to 0.2414]
Statistical Analysis 9: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Ulnar at humerus; Kendall's tau correlation coefficient = 0.1067521, 95% CI 2-sided [-0.5204 to 0.6392]
Statistical Analysis 10: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Ulnar at axilla; Kendall's tau correlation coefficient = 0.0549235, 95% CI 2-sided [-0.4633 to 0.5594]
Statistical Analysis 11: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — C6; Kendall's tau correlation coefficient = -0.2597622, 95% CI 2-sided [-0.6816 to 0.1857]
Statistical Analysis 12: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — C7; Kendall's tau correlation coefficient = -0.0129034, 95% CI 2-sided [-0.4476 to 0.4025]
Statistical Analysis 13: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by hand dynamometer; Test type: Other — Vagus; Kendall's tau correlation coefficient = 0.02457737, 95% CI 2-sided [-0.3506 to 0.4596]

8. Secondary Outcome: Strength, as Measured by Medical Research Council (MRC)
Description: The Medical Research Council (MRC) total score ranges from 0-60, with higher values indicating greater muscle strength. The MRC total score is the sum score of the following muscle group subscales (each assessed on the left side and right side): bilateral shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion. Each muscle group subscale is rated 0-5, with 0 being no movement and 5 being full strength.
Time Frame: Day 0, Day 7
Population: Participants with data collected at each time point. Not applicable to the Control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GBS Patients | Controls
Number analyzed (Participants) | 13 | 0
score on a scale
  Day 0 | 40.00 (18.64) |
  Day 7: number analyzed (Participants) | 1 | 0
  Day 7 | 56.00 (0) |
Statistical Analysis 1: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Median at wrist; Kendall's tau correlation coefficient = 0.1704986, 95% CI 2-sided [-0.3950 to 0.6584]
Statistical Analysis 2: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Median at forearm; Kendall's tau correlation coefficient = 0.1704986, 95% CI 2-sided [-0.3950 to 0.6584]
Statistical Analysis 3: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Median at cubital fossa; Kendall's tau correlation coefficient = 0.09040847, 95% CI 2-sided [-0.3821 to 0.5979]
Statistical Analysis 4: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Median at humerus; Kendall's tau correlation coefficient = 0.02501955, 95% CI 2-sided [-0.4158 to 0.4790]
Statistical Analysis 5: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Median at axilla; Kendall's tau correlation coefficient = -0.0349215, 95% CI 2-sided [-0.5033 to 0.4430]
Statistical Analysis 6: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Ulnar at wrist; Kendall's tau correlation coefficient = -0.0961, 95% CI 2-sided [-0.5458 to 0.4037]
Statistical Analysis 7: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Ulnar at forearm; Kendall's tau correlation coefficient = -0.2239171, 95% CI 2-sided [-0.6514 to 0.2935]
Statistical Analysis 8: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Ulnar at cubital fossa; Kendall's tau correlation coefficient = -0.0805076, 95% CI 2-sided [-0.5371 to 0.2974]
Statistical Analysis 9: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Ulnar at humerus; Kendall's tau correlation coefficient = 0.2910126, 95% CI 2-sided [-0.2791 to 0.7651]
Statistical Analysis 10: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Ulnar at axilla; Kendall's tau correlation coefficient = 0.02342428, 95% CI 2-sided [-0.4531 to 0.5267]
Statistical Analysis 11: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — C6; Kendall's tau correlation coefficient = 0.06536087, 95% CI 2-sided [-0.2786 to 0.4454]
Statistical Analysis 12: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — C7; Kendall's tau correlation coefficient = 0.2207792, 95% CI 2-sided [-0.2459 to 0.6708]
Statistical Analysis 13: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and strength by MRC sum score; Test type: Other — Vagus; Kendall's tau correlation coefficient = 0.14415, 95% CI 2-sided [-0.2333 to 0.4899]

9. Secondary Outcome: Number of Participants With Autonomic Dysfunction
Description: Autonomic dysfunction will be either present or absent by chart review during hospitalization.
Time Frame: During hospitalization, up to approximately 20 days
Population: Not applicable to the Control group.
Measure: Count of Participants; unit: Participants
Arm/Group | GBS Patients | Controls
Number analyzed (Participants) | 14 | 0
Participants | 5 |
Statistical Analysis 1: Comparison: GBS Patients; Null hypothesis: Nerve ultrasound measurement has no effect on the log-odds of having autonomic dysfunction (i.e., higher ultrasound measurements do not predict whether a subject has autonomic dysfunction during their hospitalization); Test type: Other — Median at wrist; p = 0.548, Regression, Logistic; Odds Ratio (OR) = 0.9310743
Statistical Analysis 2: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — Median at forearm; p = 0.548, Regression, Logistic; Odds Ratio (OR) = 0.9310743
Statistical Analysis 3: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — Median at cubital fossa; p = 0.250, Regression, Logistic; Odds Ratio (OR) = 1.23944918
Statistical Analysis 4: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — Median at humerus; p = 0.874, Regression, Logistic; Odds Ratio (OR) = 0.9613236
Statistical Analysis 5: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — Median at axilla; p = 0.698, Regression, Logistic; Odds Ratio (OR) = 0.9442314
Statistical Analysis 6: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — Ulnar at wrist; p = 0.665, Regression, Logistic; Odds Ratio (OR) = 1.193941
Statistical Analysis 7: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — Ulnar at forearm; p = 0.820, Regression, Logistic; Odds Ratio (OR) = 1.0524489
Statistical Analysis 8: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — Ulnar at cubital fossa; p = 0.193, Regression, Logistic; Odds Ratio (OR) = 1.21669122
Statistical Analysis 9: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — Ulnar at humerus; p = 0.314, Regression, Logistic; Odds Ratio (OR) = 1.2994068
Statistical Analysis 10: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — Ulnar at axilla; p = 0.405, Regression, Logistic; Odds Ratio (OR) = 1.1015629
Statistical Analysis 11: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — C6; p = 0.389, Regression, Logistic; Odds Ratio (OR) = 0.9140133
Statistical Analysis 12: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — C7; p = 0.139, Regression, Logistic; Odds Ratio (OR) = 0.7982946
Statistical Analysis 13: Comparison: GBS Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other — Vagus; p = 0.622, Regression, Logistic; Odds Ratio (OR) = 0.9330042

10. Secondary Outcome: Disability as Measured by the Guillain-Barre Syndrome (GBS) Disability Score
Description: The GBS disability score ranges from 0-6 with lower scores indicating a better outcome (0 is healthy, 6 is death).
Time Frame: Day 0, Day 7, Discharge (up to approximately 20 days), Day 90, Day 180
Population: Not applicable to the Control group. Only one participant had data collected at Day 7.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GBS Patients | Controls
Number analyzed (Participants) | 14 | 0
score on a scale
  Day 0 | 3.57 (1.02) |
  Day 7: number analyzed (Participants) | 1 | 0
  Day 7 | 3.00 (0) |
  Discharge | 3.14 (0.95) |
  Day 90 | 2.21 (1.37) |
  Day 180 | 1.64 (1.45) |
Statistical Analysis 1: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and GBS Disability score at 3 months after enrollment; Test type: Other — Median at wrist, 3 months; Kendall's tau correlation coefficient = 0.2641183, 95% CI 2-sided [-0.2344 to 0.7511]
Statistical Analysis 2: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — Median at forearm, 3 months; Kendall's tau correlation coefficient = 0.02596308, 95% CI 2-sided [-0.4859 to 0.5555]
Statistical Analysis 3: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — Median at cubital fossa, 3 months; Kendall's tau correlation coefficient = 0.05162687, 95% CI 2-sided [-0.3342 to 0.4170]
Statistical Analysis 4: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — Median at humerus, 3 months; Kendall's tau correlation coefficient = -0.1714461, 95% CI 2-sided [-0.6473 to 0.2723]
Statistical Analysis 5: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — Median at axilla, 3 months; Kendall's tau correlation coefficient = -0.0531775, 95% CI 2-sided [-0.5830 to 0.4451]
Statistical Analysis 6: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — Ulnar at wrist, 3 months; Kendall's tau correlation coefficient = 0.1371924, 95% CI 2-sided [-0.3592 to 0.6944]
Statistical Analysis 7: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — Ulnar at forearm, 3 months; Kendall's tau correlation coefficient = -0.0134595, 95% CI 2-sided [-0.5145 to 0.4627]
Statistical Analysis 8: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — Ulnar at cubital fossa, 3 months; Kendall's tau correlation coefficient = 0.01313517, 95% CI 2-sided [-0.5056 to 0.4833]
Statistical Analysis 9: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — Ulnar at humerus, 3 months; Kendall's tau correlation coefficient = -0.1196495, 95% CI 2-sided [-0.5876 to 0.3467]
Statistical Analysis 10: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — Ulnar at axilla, 3 months; Kendall's tau correlation coefficient = 0.00, 95% CI 2-sided [-0.3682 to 0.3885]
Statistical Analysis 11: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — C6, 3 months; Kendall's tau correlation coefficient = 0.1194695, 95% CI 2-sided [-0.4220 to 0.6686]
Statistical Analysis 12: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — C7, 3 months; Kendall's tau correlation coefficient = -0.0593456, 95% CI 2-sided [-0.5651 to 0.4540]
Statistical Analysis 13: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 1]; Test type: Other — Vagus, 3 months; Kendall's tau correlation coefficient = -0.1920694, 95% CI 2-sided [-0.5490 to 0.238]
Statistical Analysis 14: Comparison: GBS Patients; Null hypothesis: There is no correlation between nerve ultrasound measurements and GBS Disability score at 6 months after enrollment; Test type: Other — Median at wrist, 6 months; Kendall's tau correlation coefficient = 0.3150905
Statistical Analysis 15: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — Median at forearm, 6 months; Kendall's tau correlation coefficient = 0.1203751
Statistical Analysis 16: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — Median at cubital fossa, 6 months; Kendall's tau correlation coefficient = 0.2526605, 95% CI 2-sided [-0.1865 to 0.6430]
Statistical Analysis 17: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — Median at humerus, 6 months; Kendall's tau correlation coefficient = -0.0736010, 95% CI 2-sided [-0.5806 to 0.4223]
Statistical Analysis 18: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — Median at axilla, 6 months; Kendall's tau correlation coefficient = 0.01369735, 95% CI 2-sided [-0.5619 to 0.5236]
Statistical Analysis 19: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — Ulnar at wrist, 6 months; Kendall's tau correlation coefficient = 0.2685663, 95% CI 2-sided [-0.2488 to 0.7683]
Statistical Analysis 20: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — Ulnar at forearm, 6 months; Kendall's tau correlation coefficient = 0.1802776, 95% CI 2-sided [-0.2573 to 0.6027]
Statistical Analysis 21: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — Ulnar at cubital fossa, 6 months; Kendall's tau correlation coefficient = 0.2571327, 95% CI 2-sided [-0.2595 to 0.6227]
Statistical Analysis 22: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — Ulnar at humerus, 6 months; Kendall's tau correlation coefficient = -0.0684867, 95% CI 2-sided [-0.5757 to 0.3944]
Statistical Analysis 23: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — Ulnar at axilla, 6 months; Kendall's tau correlation coefficient = 0.1929429, 95% CI 2-sided [-0.1828 to 0.5550]
Statistical Analysis 24: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — C6, 6 months; Kendall's tau correlation coefficient = 0.1975146, 95% CI 2-sided [-0.3557 to 0.7344]
Statistical Analysis 25: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — C7, 6 months; Kendall's tau correlation coefficient = -0.0754722, 95% CI 2-sided [-0.6150 to 0.5083]
Statistical Analysis 26: Comparison: GBS Patients; [analysis description as in outcome 10, analysis 14]; Test type: Other — Vagus, 6 months; Kendall's tau correlation coefficient = -0.0706753, 95% CI 2-sided [-0.5042 to 0.3963]

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected.
Description: Adverse Events were not collected.
Arm/Group | GBS Patients | Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT04053452/Prot_001.pdf